CLINICAL TRIAL: NCT05129241
Title: Non-interventional Study on the Monthly Administration of 300 mg AliRocumab (PRALUENT®) With the 2 ml SYDNEY Auto-injector (MARS-NIS)
Brief Title: Non-interventional Study on the Monthly Administration of 300 mg AliRocumab (PRALUENT®) With the 2 ml SYDNEY Auto-injector
Acronym: MARS
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17242; U1111-1265-6221 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-11-15; First posted 2021-11-22 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Primary Hypercholesterolaemia and Mixed Dyslipidaemia; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Patients for whom the treating physician has decided to initiate lipid-lowering treatment with the PRALUENT® 2 ml SYDNEY auto-injector, irrespective of participation in the study

SUMMARY:
Primary objectives:

* To assess the effectiveness of the PRALUENT® 2 ml SYDNEY auto-injector as measured by the lipid-lowering effect of alirocumab after approx. 12 weeks treatment
* To assess the treatment satisfaction, as well as patient adherence and persistence after approximately 12 weeks of treatment with the PRALUENT® 2 ml SYDNEY auto-injector

Secondary objective:

Safety and tolerability

DETAILED DESCRIPTION:
Study duration per participant is approximately 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Primary hypercholesterolaemia (heterozygous familial or non-familial) or mixed dyslipidaemia AND confirmed vascular disease(*) AND other regular risk factors(**), OR confirmed familial heterozygous hypercholesterolaemia
* Documented maximum dietary and drug lipid-lowering therapy within the last 12 months
* Inadequate reduction of low-density lipoprotein cholesterol (LDL-C) despite maximum possible dietary and lipid-lowering therapy
* The decision of the treating physician to use the PRALUENT® 2 ml SYDNEY auto-injector regardless of study enrolment
* No previous therapy with a proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitor OR prior treatment with a PCSK9 inhibitor every 2 weeks (Q2W) or monthly (Q4W)
* Signed Informed Consent Form

(*) Coronary heart disease (CHD), cerebrovascular manifestation, peripheral arterial occlusive disease (PAOD)

(**) For cardiovascular events (e.g. diabetes mellitus, renal function glomerular filtration rate (GFR) < 60 ml/min)

Exclusion Criteria:

* Planned or existing pregnancy, cancer, drug or alcohol abuse, dementia, or general inability to understand the content of the observational study
* Existing treatment by lipid apheresis
* Age < 18 years
* Contraindications to treatment with alirocumab (PRALUENT®) according to the SmPC
* Current participation in a clinical study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary hypercholesterolaemia (heterozygous familial and non-familial) or mixed dyslipidaemia and confirmed cardiovascular disease and with regular additional risk factors, and/or patients with confirmed familial heterozygous hypercholesterolaemia for whom the treating physician has decided to initiate lipid-lowering treatment with the PRALUENT® 2 ml SYDNEY auto-injector, irrespective of participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline to week 12 in low-density lipoprotein cholesterol (LDL-C) | from baseline to week 12
Percent change from baseline to week 12 in low-density lipoprotein cholesterol (LDL-C) | from baseline to week 12
Treatment acceptance assessed using the Injection Treatment Acceptance Questionnaire (ITAQ) | week 12

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 12 weeks
Number of quality defects assessed using product complaints | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number, Germany, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Parhofer KG, Bramlage P, Gries C, Harder C, Look C, Paar WD, Rauch-Krohnert U. Lipid-Lowering Efficiency and Safety of Alirocumab 300 mg Using a 2-mL Autoinjector Device in Real-World Practice: The MARS Study. Drugs Real World Outcomes. 2025 Mar;12(1):63-74. doi: 10.1007/s40801-024-00471-w. Epub 2025 Jan 28. PMID 39875772